CLINICAL TRIAL: NCT01423916
Title: A Parallel-arm, Double-blind, Placebo and Positive Controlled Multiple Oral Dose Administration Trial to Evaluate the Effects of OPC-34712 on QT/QTc in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Trial to Evaluate the Effects of OPC-34712 on QT/QTc in Subjects With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-10-242
Record Dates: First submitted 2011-08-08; First posted 2011-08-26 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; QTc Interval
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (OPC-34712, placebo) (Active Comparator): Arm 1 will be administered 4 mg OPC-34712 once daily (QD) for 11 days and OPC-34712 placebo for 1 day.
  Interventions: Drug: OPC-34712 (4mg); Drug: Placebo
- Arm 2 (OPC-34712, placebo) (Active Comparator): Arm 2 will be administered 12 mg OPC-34712 QD for 11 days and OPC-34712 placebo for 1 day.
  Interventions: Drug: OPC-34712 (12mg); Drug: Placebo
- Arm 3 (moxifloxacin, placebo) (Active Comparator): Arm 3 will be administered 400 mg moxifloxacin (positive control) plus OPC-34712 placebo for 1 day and OPC-34712 placebo QD for 11 days.
  Interventions: Drug: Moxifloxacin; Drug: Placebo
- Arm 4 (moxifloxacin, placebo) (Active Comparator): Arm 4 will be administered OPC-34712 placebo QD for 11 days and 400 mg moxifloxacin (positive control) plus OPC-34712 placebo for one day.
  Interventions: Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: OPC-34712 (4mg) — Arms assigned to this intervention receive 4mg.
  Arms: Arm 1 (OPC-34712, placebo)
Drug: Moxifloxacin — Arms assigned to this intervention will receive 400mg.
  Arms: Arm 3 (moxifloxacin, placebo); Arm 4 (moxifloxacin, placebo)
Drug: OPC-34712 (12mg) — Arms assigned to this intervention receive 12mg.
  Arms: Arm 2 (OPC-34712, placebo)
Drug: Placebo — OPC-34712 placebo

SUMMARY:
The purpose of this study is to establish pharmacodynamics (PD), pharmacokinetics (PK), and adverse event (AE) profile of OPC-34712 administered to schizophrenic/schizoaffective subjects. The goals of this trial are three-fold:

* To determine the effect of OPC-34712 on the individual QT interval (QTcI) corrected for placebo
* To determine the effect of moxifloxacin on QTcI
* To examine the concentration-effect relationship of OPC-34712 and moxifloxacin on QTcI

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 55 years of age, inclusive, with a diagnosis of schizophrenia or schizoaffective disorder as defined by DSM-IV-TR criteria.
* Body mass index of 19 to 35 kg/m2.

Exclusion Criteria:

* Females who are pregnant or lactating. A negative serum pregnancy test must be confirmed prior to the first dose of trial medication for all female subjects.
* Subjects presenting with a first episode of schizophrenia or schizoaffective disorder based on the clinical judgment of the investigator.
* Subjects who have received continuous medication therapy to treat schizophrenia or schizoaffective disorder for less than 6 months prior to washout.
* Subjects with schizophrenia or schizoaffective disorder that are considered resistant/refractory to antipsychotic treatment by history, who have a history of failure to clozapine, or who are responsive only to clozapine treatment.
* Subjects with a current DSM-IV-TR Axis I diagnosis other than schizophrenia or schizoaffective disorder.
* Hospitalization for an exacerbation of schizophrenia or schizoaffective disorder within 3 months prior to randomization.
* Subjects who have a history of or who have evidence of other medical and/or neurological conditions that would expose them to an undue risk of a significant AE or interfere with assessments of safety or efficacy during the course of the trial.
* Subjects with a history of neuroleptic malignant syndrome.
* Subjects with a history of seizure disorder.
* Subjects who meet DSM-IV-TR criteria for substance dependence within 6 months prior to randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Otsuka Investigational Site, Long Beach, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site, Fort Lauderdale, Florida
  - Otsuka Investigational Site, Overland Park, Kansas
  - Otsuka Investigational Site, Rockville, Maryland
  - Otsuka Investigational Site, St Louis, Missouri
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, placebo and positive-controlled, parallel-arm study to examine the effects of 2 dose levels of brexpiprazole on the QT/QTc (QT interval corrected for heart rate) interval. This study was run in 8 sites in the US.
Pre-assignment Details: Participants were screened from Days -28 to -6 and washed out from their current antipsychotic medication between Days -5 to -2 and resumed antipsychotic therapy by study physician on Day 13 or at early termination (ET). A safety Follow-up was done 30 (+2) days after last dose of study medication.
Groups:
- Brexpiprazole 4mg: Participants received 4mg brexpiprazole (as four 1-mg tablets) QD (once daily) on Days 1 to 11 and brexpiprazole placebo (as 4 tablets) QD on Day 12.
- Brexpiprazole 12mg: Participants received 12mg brexpiprazole (as two 5-mg tablets and two 1-mg tablets) QD on Days 1 to 11 and brexpiprazole placebo (as 4 tablets) QD on Day 12.
- Moxifloxacin/Placebo: Moxifloxacin/Placebo arm comprised of 2 groups: one who had received 400 mg moxifloxacin (as 1 tablet) plus brexpiprazole placebo (as 3 tablets) on Day 1 and brexpiprazole placebo (as 4 tablets) QD on Days 2 to 12 and the other group who received brexpiprazole placebo (as 4 tablets) QD on Days 1 to 11 and 400 mg moxifloxacin (as 1 tablet) plus brexpiprazole placebo (as 3 tablets) on Day 12.
Period: Overall Study
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin/Placebo
Started | 74 | 73 | 71
Completed | 63 | 53 | 64
Not Completed | 11 | 20 | 7
Not completed — Adverse Event | 5 | 9 | 2
Not completed — Met Withdrawal Criteria | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 10 | 3
Not completed — Protocol Deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole 4mg: Participants received 4mg brexpiprazole (as four 1-mg tablets) QD on Days 1 to 11 and brexpiprazole placebo (as 4 tablets) QD on Day 12.
- Brexpiprzole 12mg: Participants received 12mg brexpiprazole (as two 5-mg tablets and two 1-mg tablets) QD on Days 1 to 11 and brexpiprazole placebo (as 4 tablets) QD on Day 12.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 4mg | Brexpiprzole 12mg | Moxifloxacin/Placebo | Total
Number analyzed (Participants) | 74 | 73 | 71 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (9.6) | 37.5 (9.0) | 38.2 (9.6) | 38.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 15 | 49
  Male | 56 | 57 | 56 | 169

OUTCOME MEASURES:

1. Primary Outcome: Time-matched QTcI Change From Baseline (Day -1) Corrected for Placebo on Day 11 Following Brexpiprazole Treatment.
Description: Pharmacodynamics endpoint is the time-matched corrected QT interval (QTcI) change from baseline (Day -1) corrected for placebo on Day 11 following brexpiprazole treatment. The primary QT to QTc correction formula (QTcI) was determined for each participant using the participant's baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k was derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k).
Time Frame: Day 11 (Hours 1, 2, 3, 4, 5, 6, 8, 12, 16, 24)
Population: The dataset quantitates effect of brexpiprazole on individual QTcI corrected for placebo of the completer population where participants received study medication from Day 1 to Day 11 (placebo at Day 1) had 1 Predose and Post-dose time-matched ECG assessments on Day 1 and Day 11. The first 5 time points for moxifloxacin arm only were 2-sided 98% CI.
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Moxifloxacin/Placebo | Brexpiprazole 12mg | Brexpiprazole 4mg
Number analyzed (Participants) | 64 | 53 | 63
msec
  Hours 1 (N=61, 53, 61) | 9.2 [5.8 to 12.6] | -0.2 [-5.2 to 4.8] | 2.6 [-2.2 to 7.4]
  Hours 2 (N= 62, 53, 62) | 9.4 [6.0 to 12.8] | -0.2 [-5.0 to 4.5] | 1.2 [-3.4 to 5.7]
  Hours 3 (N= 60, 51, 61) | 8.5 [5.1 to 11.9] | 1.3 [-3.4 to 6.0] | 1.1 [-3.4 to 5.6]
  Hours 4 (N= 62, 53, 62) | 10.5 [7.1 to 13.8] | 3.1 [-1.7 to 8.0] | 3.6 [-1.0 to 8.3]
  Hours 5 (N= 62, 52, 62) | 6.2 [2.8 to 9.5] | -0.2 [-5.1 to 4.6] | 1.7 [-2.9 to 6.3]
  Hours 6 (N= 61, 52, 62) | 7.3 [3.8 to 10.7] | 1.3 [-3.5 to 6.1] | 8.3 [-3.7 to 12.9]
  Hours 8 (N= 59, 50, 59) | 7.5 [4.1 to 10.9] | 2.5 [-2.0 to 6.9] | 4.0 [-0.2 to 8.3]
  Hours 10 (N= 59, 47, 56) | 9.0 [5.5 to 12.4] | 2.2 [-2.3 to 6.8] | 5.2 [0.8 to 9.5]
  Hours 12 (N= 58, 47, 58) | 6.8 [3.3 to 10.3] | 2.6 [-2.2 to 7.4] | 5.3 [0.7 to 9.9]
  Hours 16 (N= 59, 48, 53) | 2.2 [-1.3 to 5.7] | 0.8 [-3.9 to 5.5] | 4.0 [-0.6 to 8.5]
  Hours 24 (N= 54, 45, 57) | 2.1 [-1.5 to 5.7] | 0.7 [-4.2 to 5.7] | 0.1 [-4.6 to 4.8]

2. Primary Outcome: Number of Participants With Adverse Events (AE) and Clinically Important Changes in Vital Signs, Physical Examinations, Laboratory Tests, and Standard ECGs (Electrocardiogram).
Description: Clinically important changes in vital signs, physical examinations, laboratory tests and ECGs were by and large reflected in AE/SAE (which are presented in safety section) of this report.
Time Frame: AEs were recorded from Screening (informed consent was signed) during the 12-day treatment period to follow-up 30 (+ 2) days post-last dose of study medication
Population: Safety dataset of randomized participants received 1 dose of study medication after Day 1.
Measure: Number; unit: participants
Groups:
- Moxifloxacin: Moxifloxacin arm comprised of all participants who had received 400 mg moxifloxacin (as 1 tablet) on Day 1 and Day 12.
- Placebo: Placebo arm comprised of all participants who received brexpiprazole placebo (as 3 tablets) on Day 1 and as 4 tablets QD on Days 2 to 12; and brexpiprazole placebo (as 4 tablets) QD on Days 1 to 11 and as 3 tablets on Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 70 | 67 | 65 | 68
participants
  Postural orthostatic tachycardia syndrome | 0 | 1 | 0 | 0
  Tachycardia | 0 | 0 | 2 | 1
  Blood creatinine phosphokinase increased | 1 | 1 | 0 | 0
  Blood pressure increased | 0 | 0 | 0 | 1
  Blood prolactin increased | 0 | 0 | 1 | 0
  Hepatic enzyme increased | 1 | 1 | 0 | 0
  Liver function test abnormal | 0 | 1 | 0 | 0
  Weight increased | 0 | 1 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0

3. Primary Outcome: Maximum Peak Plasma Concentration (Cmax) of Brexpiprazole and Moxifloxacin.
Description: Pharmacokinetics endpoint is the maximum (peak) plasma concentration (Cmax) of brexpiprazole and moxifloxacin. Values for Cmax were determined directly from the observed data. Blood samples were collected on Days -1, 1, 11, and 12 at predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose or at ET.
Time Frame: Day 11
Population: Pharmacokinetics (PK) analysis dataset consisted of all evaluable PK parameters from randomized participants who had plasma concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Moxifloxacin/ Placebo: Moxifloxacin/Placebo arm comprised of 2 groups: one who had received 400 mg moxifloxacin (as 1 tablet) plus brexpiprazole placebo (as 3 tablets) on Day 1 and brexpiprazole placebo (as 4 tablets) QD on Days 2 to 12 and the other group who received brexpiprazole placebo (as 4 tablets) QD on Days 1 to 11 and 400 mg moxifloxacin (as 1 tablet) plus brexpiprazole placebo (as 3 tablets) on Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin/ Placebo
Number analyzed (Participants) | 63 | 53 | 64
ng/mL | 170 (69.8) | 462 (249) | 2760 (659)

4. Primary Outcome: Time to Maximum (Peak) Plasma Concentration (Tmax) of Brexpiprazole and Moxifloxacin.
Description: Pharmacokinetics endpoint is the time to maximum (peak) plasma concentration (tmax) of brexpiprazole and moxifloxacin. Values for tmax were determined directly from the observed data. Blood samples were collected on Days -1, 1, 11, and 12 at predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose or at ET.
Time Frame: Day 11
Population: PK analysis dataset consisted of all evaluable PK parameters from randomized participants who had plasma concentrations.
Measure: Median (Full Range); unit: Hours
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin/ Placebo
Number analyzed (Participants) | 63 | 53 | 64
Hours | 3.54 [1.00 to 8.00] | 3.00 [0.00 to 8.00] | 1.25 [0.00 to 5.00]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve During Dosing (AUCT).
Description: Pharmacokinetics endpoint is the area under the concentration-time curve from time zero to 24 hours (AUC0-24h) of brexpiprazole and moxifloxacin. Area under the plasma concentration-time curve during the dosing interval at steady-state (AUCT) value was estimated using the linear trapezoidal rule; the value reported represent the area under the curves to the last time point during that day. Blood samples were collected on Days -1, 1, 11, and 12 at predose, and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose or at ET.
Time Frame: Day 11
Population: PK analysis dataset consisted of all evaluable PK parameters from randomized participants who had plasma concentrations. For Moxifloxacin group, area under the plasma concentration-time curve was calculated to the last observable concentration.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin/ Placebo
Number analyzed (Participants) | 63 | 53 | 64
ng*h/mL | 3100 (1400) | 8880 (5110) | 28400 (6350)

6. Secondary Outcome: Number of Participants Noted With Time-matched Change in Mean QTcI Change From Baseline for Assay Sensitivity of Moxifloxacin Treatment Corrected for Placebo at Day 11.
Description: New onset (> 450, > 480, or > 500 msec) in QTc was defined as a participant who attained a QTc > 450, > 480, > 500 msec during Day 11 but not on Day -1. The number of participants were noted with time-matched change in mean QTcI change from Baseline for assay sensitivity of moxifloxacin treatment corrected for placebo. The primary QT to QTc correction formula (QTcI) were determined for each participant using the participant's Baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k were derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k).
Time Frame: Baseline, Day 11
Population: Assay sensitivity dataset demonstrated the effect of moxifloxacin on QTcI from randomized participants in moxifloxacin and placebo arms who had evaluable time-matched ECG assessments on Days -1, 1, 11, and 12. Number of participants analyzed included those who had observations in QTc at both Days -1 and 11.
Measure: Number; unit: participants
Groups:
- Moxifloxacin 400 mg: Moxifloxacin arm comprised of all participants who had received 400 mg moxifloxacin (as 1 tablet) on Day 1 and Day 12.
- Placebo: Placebo arm comprised of all participants who had received brexpiprazole placebo (as 3 tablets) on Day 1 and as 4 tablets QD on Days 2 to 12; and brexpiprazole placebo (as 4 tablets) QD on Days 1 to 11 and as 3 tablets on Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants
  QTcI (> 450 msec) | 5 | 4 | 5 | 0
  QTcI (> 480 msec) | 0 | 1 | 0 | 0
  QTcI (> 500 msec) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Summary of Maximum QTcI on Day 11 Minus Mean QTcI on Day -1 (Baseline).
Description: The primary QT to QTc correction formula (QTcI) were determined for each participant using the participant's Baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k were derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k). The change form Baseline in summary of maximun QTcI on Day 11 minus mean QTcI on Day -1 (Baseline) is presented here.
Time Frame: Baseline, Day 11
Population: Assay sensitivity dataset shows the effect of moxifloxacin on QTcI from randomized participants in moxifloxacin and placebo arms who had evaluable time-matched ECG assessments on Days -1, 1, 11, and 12. Number of participants analyzed were total number of participants with both Baseline and at least one observation of the given parameter.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Moxifloxacin 400mg: Moxifloxacin arm comprised of all participants who had received 400 mg moxifloxacin (as 1 tablet) on Day 1 and Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 62 | 62
msec | 11.6 (7.4) | 12.4 (10.4) | 10.6 (7.7) | -1.1 (13.1)

8. Secondary Outcome: Change From Baseline in Summary of Maximum QTcI on Day 11 Minus Maximum QTcI on Day -1 (Baseline).
Description: The primary QT to QTc correction formula (QTcI) were determined for each participant using the participant's Baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k were derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k). The change from Baseline in summary of maximum QTcI on Day 11 minus maximum QTcI on Day -1 (Baseline) is presented here.
Time Frame: Baseline, Day 11
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Moxifloaxcin 400mg: Moxifloxacin arm comprised of all participants who had received 400 mg moxifloxacin (as 1 tablet) on Day 1 and Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloaxcin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 62 | 62
msec | 0.4 (9.1) | 0.9 (10.9) | 0.0 (8.1) | -1.2 (8.0)

9. Secondary Outcome: Number of Participants With QTcI Interval Between 30 and 60 Msec on Day 11.
Description: The primary QT to QTc correction formula (QTcI) were determined for each participant using the participant's Baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k were derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k). Participants with QTcI interval change between 30 to 60 msec were presented here.
Time Frame: Day 11
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants | 4 | 1 | 11 | 2

10. Secondary Outcome: Number of Participants With QTcI Interval > 60 Msec on Day 11.
Description: The primary QT to QTc correction formula (QTcI) were determined for each participant using the participant's Baseline (Day -1 placebo) ECG data. The QT correction formula QT / (RR)k were derived using log-log-linear regression, where log (QT) = a + k × log (RR) + ε to estimate the exponent (k). Participants with QTcI interval change of > 60 msec on Day 11 were presented here.
Time Frame: Day 11
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number Participants Noted With New Incidence of QT Interval of > 500 Msec on Day 11.
Description: The number of participants who were noted with new incidence of QT interval of > 500 msec on Day 11 and a 12-lead ECG was used.
Time Frame: Day 11
Population: Assay sensitivity sample dataset demonstrated the ability of the trial that detected the effect of moxifloxacin on the QTcI that consisted from randomized participants in moxifloxacin and placebo arms, who had evaluable time-matched ECG assessments in both periods (Day -1/1 or Day 11/12) in placebo and moxifloxacin on Days -1, 1, 11, and 12.
Measure: Number; unit: participants
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With New Incidence of ECG Morphology Abnormalities on Day 11.
Description: Participants with incidence of ECG morphology abnormalities on Day 11 (participants who had abnormalities during Day 11 but not at Day -1) were noted. Types of abnormalities included appearance of abnormal U waves, negative T waves, elevation of ST segment, depression of ST segment, second degree heart block, third degree heart block, right bundle branch block, and left bundle branch block. ECGs were sampled at predose and approximately 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose on Days -1, 1, 11, and 12.
Time Frame: Day 11
Population: Number of participants who took at least one dose of study drug post Day -1, and had evaluations of the ECG parameters at Baseline and Post Baseline.
Measure: Number; unit: participants
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants
  U Wave abnormalities | 0 | 0 | 0 | 0
  Negative T Waves | 4 | 7 | 8 | 6
  Depression of ST segment | 2 | 2 | 4 | 1
  Elevation of ST segment | 0 | 0 | 0 | 0
  Second degree heart block | 0 | 0 | 0 | 0
  Third degree heart block | 0 | 0 | 0 | 0
  Right bundle branch block | 0 | 0 | 0 | 0
  Left bundle branch block | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Maximum Change From Baseline to the On-treatment ECG Values on Day 11 for Heart Rate (HR), PR Interval, and QRS Interval.
Description: Changes in HR with values 25% decrease from Day -1 and HR < 50 bpm and 25% increase from Day -1 and HR > 100 bpm; PR interval of greater than or equal to 25% change from Day -1 and PR > 200 msec; QRS interval of Greater than or equal to 25% change from Day -1 and > 100 msec were noted on Day 11. Maximum change from baseline to the on-treatment ECG values on Day 11 for heart rate.
Time Frame: Day 11
Population: Electrocardiograms were sampled at predose and approximately 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose on Days -1, 1, 11, and 12.
Measure: Number; unit: participants
Groups:
- Brexpiprazole 4mg: Participants were randomised to 1 of 4 arms in a ratio of 2:2:1:1. On Day 1, all participants received brexpiprazole placebo tablets. Participants received 4mg brexpiprazole (as four 1-mg tablets) QD on Days 1 to 11 and brexpiprazole placebo (as 4 tablets) QD on Day 12.
- Brexpiprazole 12mg: Participants were randomised to 1 of 4 arms in a ratio of 2:2:1:1. On Day 1, all participants received brexpiprazole placebo tablets. Participants received 12mg brexpiprazole (as two 5-mg tablets and two 1-mg tablets) and brexpiprazole placebo (as 4 tablets) QD on Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 62 | 53 | 63 | 62
participants
  HR: < 50 bpm | 0 | 0 | 0 | 0
  HR: > 100 bpm | 5 | 7 | 2 | 4
  PR > 200 msec | 0 | 0 | 0 | 0
  QRS > 100 msec | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were recorded from Screening (informed consent was signed) throughout the 12-day treatment period until follow-up of up to 30 (+ 2) days post-last dose of study medication.
Description: The safety dataset consisted of all randomized participants who had received at least 1 oral dose of study medication after Baseline (Day 1) to Day 12.
Arm/Group | Brexpiprazole 4mg | Brexpiprazole 12mg | Moxifloxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/67 | 0/65 | 0/68
Other Adverse Events (participants affected / at risk) | 27/70 | 27/67 | 9/65 | 20/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 4mg (N=70) | Brexpiprazole 12mg (N=67) | Moxifloxacin (N=65) | Placebo (N=68)
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 4mg (N=70) | Brexpiprazole 12mg (N=67) | Moxifloxacin (N=65) | Placebo (N=68)
Constipation (Gastrointestinal disorders) | 3 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 5 | 1 | 4
Application site dermatitis (General disorders) | 6 | 1 | 2 | 4
Akathisia (Nervous system disorders) | 5 | 5 | 1 | 1
Dizziness (Nervous system disorders) | 6 | 8 | 2 | 1
Extrapyramidal disorder (Nervous system disorders) | 4 | 5 | 0 | 1
Somnolence (Nervous system disorders) | 3 | 4 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 4 | 0 | 3
Restlessness (Psychiatric disorders) | 2 | 5 | 0 | 3
Headache (Nervous system disorders) | 1 | 5 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No